CLINICAL TRIAL: NCT03529136
Title: A Prospective Multicenter Clinical Study to Evaluate The Safety and Efficiency of Human Umbilical Cord Mesenchymal Stem Cell Transfusion in Patients With Decompensated Liver Cirrhosis.
Brief Title: Clinical Trial of Umbilical Cord Mesenchymal Stem Cell Transfusion in Decompensated Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); First Affiliated Hospital of Fujian Medical University (Other); Yantai Hospital for Infectious Diseases (Unknown); The Second Affiliated Hospital of Chongqing Medical University (Other); Jinan Hospital for Infectious Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTR1800015304
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-03

CONDITIONS: Decompensated Liver Cirrhosis
Keywords: Mesenchymal Stem Cell; MSC

STUDY DESIGN:
Intervention Model Description: Patients with decompensated liver cirrhosis are going to be assigned to receive standard medical care plus UC-MSC treatment with two different protocol (group 1 and group 2) or standard medical care (control). Four times of MSC infusion (1.5x10E6 cells/kg body weight) via peripheral vein will be given to the group 1（once every 4 days), and two times of MSC infusion once every 7 days to group 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSC group 1 (Experimental): Procedure:UC-MSC infusion via peripheral vein. Four times of MSC infusion (1.5x10E6 cells/kg body weight) via peripheral vein will be given to the group 1(once every 4 days).
  Interventions: Biological: UC-MSC
- MSC group 2 (Experimental): Procedure:UC-MSC infusion via peripheral vein. Two times of MSC infusion (1.5x10E6 cells/kg body weight) via peripheral vein will be given to the group 2(once every 7 days).
  Interventions: Biological: UC-MSC
- Control group (Experimental): Control group with standard medical care. UC-MSC infusion could be considering in this group after 24 weeks' followed-up.
  Interventions: Biological: UC-MSC

INTERVENTIONS:
Biological: UC-MSC — Human umbilical cord mesenchymal stem cells have driven from Wharton's jelly and cultured with serum-free medium in Shandong Cell and tissue bank. All of the cells in this study within three passages. Before transfusion, the mesenchymal stem cells were subjected to quality control. The UC-MSC were stained with anti-CD90-FITC, Anti-CD44-FITC, Anti-CD34-FITC and anti-45-FITC.
  Other Names: Human umbilical cord mesenchymal stem cells

SUMMARY:
Decompensated liver cirrhosis is one of the life-threatening complication of chronic liver disease. Liver transplantation currently is the only effective method that can improve the survival of these patients. However, the severe shortage of donor livers, high cost, and potential serious complications have restricted the availability of liver transplantation.Umbilical cord mesenchymal stem cells (UC-MSC) has been generally shown to be safe and effective for liver diseases in some pre-clinical and clinical studies. This study aim to evaluate the safety and efficiency of human umbilical cord mesenchymal stem cell transfusion in patients with decompensated liver cirrhosis, and explore the best protocol of MSC transfusion.

DETAILED DESCRIPTION:
This study is a multicenter non randomized control study. Patients with decompensated liver cirrhosis are going to be assigned to receive standard medical care plus UC-MSC treatment with two different protocol (group 1 and group 2) or standard medical care (control). Four times of MSC infusion (1.5x10E6 cells/kg body weight) via peripheral vein will be given to the group 1（once every 4 days), and two times of MSC infusion once every 7 days to the group 2. The primary outcome is survival rates in one year. Secondary outcomes are liver function, liver ascites and MELD score.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed as decompensated liver cirrhosis.
2. Hepatitis B/C Liver Cirrhosis After Viral Treatment, HBV/HCV Viral Loads Below Detection Level over six mouths, and the liver function remained below Child-pugh A grade or MELD score >10.
3. Other causes of cirrhosis, liver function compensatory incomplete.
4. In the past year, despite active medical treatment taken, the condition has continued to increase, at least because of cirrhosis complications such as ascites, spontaneous peritonitis, gastrointestinal bleeding, and hepatic encephalopathy in hospital over one time.
5. Need to intermittently supplement albumin and apply diuretic therapy.
6. Albumin <35 g/L, total bilirubin <170 umol/L, prothrombin activity> 30%; (Prothrombin time <20 s, moderate or lower mass ascites, spontaneous peritonitis and hepatic encephalopathy (grade II or lower), Child-pugh score> 5 points).
7. There was no history of gastrointestinal hemorrhage within the last month and population with no high-risk portal hypertension and gastrointestinal bleeding was evaluated recently.
8. Unconditional acceptance of orthotopic liver transplantation.
9. Aged from 18 to 65 years.
10. Voluntarily signed informed consent form.

Exclusion Criteria:

1. A malignant tumor with liver or other organs or a history of previous cancer.
2. Complications include gastrointestinal bleeding, spontaneous peritonitis, hepatic encephalopathy, hepatorenal syndrome, and Acute infection episodes.
3. Patients with severe heart, lung, kidney or blood system diseases and failure status.
4. Pregnant or lactating women.
5. Allergic constitution.
6. There is a history of alcohol abuse, drug abuse, and failure to effectively quit. 7. Patients did not participate in other clinical trials within 4 weeks.

8. Any condition, investigator believe that patients should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | one year
  The overall survival ratio of three groups will be detection after infusion in one year.

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Wang, Principal Investigator — Jinan Hospital for Infectious Diseases